CLINICAL TRIAL: NCT05835037
Title: Clinical and Nutrigenetic Assessment of Zinc in Participants With Prediabetes
Brief Title: Effect of Zinc on Glucose Homeostasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Joshua Lewis, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HP-00105493
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prediabetic State; Hyperglycemia
MeSH Terms: conditions — Prediabetic State; Hyperglycemia | interventions — gluconic acid

STUDY DESIGN:
Intervention Model Description: Two hundred prediabetic individuals will be enrolled. The investigators will prospectively evaluate the impact of zinc supplementation on fasting glucose levels and HbA1c, through the completion of randomized, placebo-controlled study of zinc gluconate (one 30 mg tablet per day for 1 year) and placebo (1 tablet per day for 1 year). Participants will be randomized 1:1 to either zinc or placebo.
Who Masked: Participant, Care Provider
Masking Description: Enrolled subjects will be randomized (1:1) to either the zinc or placebo intervention. Clinical staff and participants will be blinded to treatment assignment. Sealed, opaque assignment envelopes will be shuffled prior to study initiation and opened sequentially by a designated member of the research team who will then deliver the correct study drug to the clinical staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc treatment (Experimental): Research subjects administered zinc gluconate for 1 year (one 30 mg tablet per day)
  Interventions: Drug: Zinc Gluconate 30 MG
- Placebo (Placebo Comparator): Research subjects administered placebo for 1 year (1 tablet per day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc Gluconate 30 MG — Participants will take one tablet per day (30 mg Zinc gluconate) for 1 year
  Arms: Zinc treatment
Drug: Placebo — Participants will take one placebo tablet per day for 1 year
  Arms: Placebo

SUMMARY:
The purpose of this investigation is to evaluate the impact of zinc supplementation on fasting glucose levels, hemoglobin A1c (HbA1c), and other indices of glucose homeostasis in individuals with prediabetes. The investigators hypothesize that prediabetic subjects receiving zinc will demonstrate a greater decrease in HbA1c and blood glucose compared to prediabetic subjects receiving placebo.

Specific Aim: Conduct a prospective, double-blind randomized clinical trial comparing the effects of 12 months of zinc supplementation (zinc gluconate 30 milligram [mg] per day) versus placebo on glucose homeostasis. Based upon expected effect size and power calculations, and anticipating a 20% drop-out rate, the investigators will study 200 prediabetic subjects (100 per group) using a 1:1 randomization design. HbA1c, fasting plasma glucose, and other measures will be obtained at 0, 6, and 12 months and will be compared between zinc supplementation and placebo groups.

DETAILED DESCRIPTION:
Subjects: 200 prediabetic, but otherwise healthy, subjects will be recruited at the Amish Research Clinic in Lancaster, PA. Recruitment of individuals with prediabetes will be facilitated through prior measurements of HbA1c (5.7 to 6.4%), or fasting blood glucose levels (100 to 125 mg/dL) if HbA1c is unavailable for a given participant, and current prediabetes status will be confirmed during eligibility screening.

Study Design and Intervention: 200 prediabetic subjects will be randomized 1:1 to either zinc gluconate (30 mg/day by mouth) or placebo for 12 months. Zinc dose and duration were selected based on available literature to maximize glucose-lowering potential and to achieve a durable effect. Eligible subjects (prediabetic men or women 18 to 80 years old) will undergo a thorough medical history, physical examination, must be able to willingly and safely discontinue all zinc-containing vitamins/supplements for at least 2 weeks prior to protocol initiation. After eligibility is established and informed consent is obtained, measures of blood and urine zinc concentration, glucose homeostasis (i.e. fasting glucose, HbA1c, insulin levels, 2h OGTT), and serum lipids will be measured at baseline (Clinic Visit #1), 6 months after treatment (Clinic Visit #2), and at 12 months of treatment (Clinic Visit #3). Samples will be banked at all 3 time points for measures of insulin processing (P:I ratio), insulin clearance (C:I ratio), and insulin sensitivity (Matsuda Index).

* Home visit to screen for eligibility: A research nurse and an Amish community liaison will visit potential research subjects in their homes. The nurse will explain the study and obtain informed consent. If a research subject consents, the nurse will obtain a medical history and screening laboratory tests to confirm prediabetes status (HbA1c = 5.7 to 6.4%) and assess eligibility (e.g. complete blood count [CBC], comprehensive metabolic panel [CMP], TSH). Participants will be excluded if they are pregnant, currently breastfeeding, have history of severe gastrointestinal (GI) disorders, upper GI surgery, hemochromatosis, cancer, liver disease, kidney disease, inadequately treated thyroid disease, or cardiovascular disease, hemoglobin < 12.5 g/dl (male) or < 11 g/dl (female), are taking medications that adversely affect glucose homeostasis (e.g., corticosteroids, anti-psychotic agents), hypersensitive to zinc, use of denture adhesive containing zinc, taking vitamins or other supplements and is unwilling or cannot safely, in the opinion of the study physician, discontinue their use at least 2 week prior to protocol initiation, or any other condition that would, in the opinion of the investigator, place them at an unacceptable risk or render them unable to meet the requirements of the protocol.
* Study Drug and Randomization: Subjects will be dispensed 190 zinc gluconate 30 mg capsules or placebo at Clinic Visit #1 and will receive additional 190 tablets after 6 months when reporting for Clinic Visit #2. Participants will be instructed to take one tablet per day at least one hour before or two hours after breakfast. A matching placebo will be developed at the Applied Pharmaceutics Laboratory at the University of Maryland School of Pharmacy. Enrolled subjects will be randomized (1:1) to either the zinc or placebo intervention. Clinical staff and participants will be blinded to treatment assignment. Sealed, opaque assignment envelopes will be shuffled prior to study initiation and opened sequentially by a designated member of the research team who will then deliver the correct study drug to the clinical staff.
* Clinic Visit #1 (baseline assessment): After collection of a first morning void urine sample for measurement of zinc levels, research subjects will be transported to the Amish Research Clinic after an overnight fast where heights, weights, and vital signs will be measured. Women of child-bearing age will undergo a pregnancy test. A brief medical history including mediation usage will be performed and a food frequency questionnaire will be administered to estimate dietary zinc intake. A catheter will be placed, and fasting blood samples will be obtained to assess zinc levels, blood glucose, HbA1c, circulating lipid levels (e.g. LDL, HDL, and triglycerides), ceruloplasmin (to monitor copper deficiency), and for sample banking. A 2h (75g) OGTT will also be performed as described below. Participants will be given a 6-month supply of zinc or placebo tablets and a logbook that they will complete throughout the study, which will document daily administration of the tablets as well as any reasons for missed doses. Adherence will be assessed by comparison of remaining pill count to logbook entry.
* Clinic Visit #2 (6 month assessment): At 6 months ± 1 week after initiation of study drug, subjects will return to the Amish Research Clinic to assess intervention compliance, changes in medication/vitamin usage, and potential adverse side effects. An identical medical exam and food frequency questionnaire will be administered, and women of child-bearing age will undergo another pregnancy test. First void urine and fasting blood samples will be collected for measurement of urinary and blood zinc levels, blood glucose, HbA1c, lipid levels, ceruloplasmin, CBC, CMP, and sample banking as described above. A 2h (75g) OGTT will also be performed. Pill count and participant logbook will be reviewed to assess adherence. Participants will receive 190 zinc or placebo tablets for use in the following 6 months and instructions regarding how and when to take them will be repeated.
* Clinic Vist #3 (12 month assessment): At 12 months ± 1 week after initiation of study drug, subjects will again return to the Amish Research Clinic. Clinic Visit #3 will be identical to Clinic Visit #2 with regards to sample collection, data capture, and methodological procedures. Logbooks and remaining tablets will be collected from each participant to assess intervention adherence.

Laboratory and Other Research Methods: Our research team routinely performs all of the clinical research methodologies and statistical analyses proposed in this clinical trial. We do not anticipate any problems executing this clinical trial within the time frame of the proposed grant period.

* Routine Laboratory Testing: Eligibility screening laboratory tests (HbA1c, CBC, CMP, TSH) and other testing (blood and urine zinc levels, fasting glucose, lipid profile, ceruloplasmin) will be performed through Quest Diagnostics. Urine pregnancy tests will be administered by Amish Research Clinic staff.
* Immunoassays: Insulin, proinsulin, and C-peptide levels will be measured by immunoassay by the Cytokine Core Laboratory of the Center for Innovative Biomedical Resources (CIBR) located at the University of Maryland, Baltimore. Standard kits, reagents and protocols will be used. To minimize inter-assay variation, all immunoassays will be batched and run after samples for the entire cohort have been collected.
* 2h Oral Glucose Tolerance Test: After an overnight fast, subjects will report to the Amish Research Clinic. An indwelling cannula will be placed in an arm vein for serial blood draws at 0, 30, 60, 90, and 120 min after administration of a glucose solution (75 g glucose in 237ml), ingested over 5 min.

ELIGIBILITY:
Inclusion Criteria:

* Amish men or women who are 18 to 80 years old
* Prediabetes (HgbA1c = 5.7-6.4% or fasting glucose levels 100-125 mg/dL)

Exclusion Criteria:

* Pregnant
* Currently breastfeeding
* History of severe gastrointestinal disorders or upper gastrointestinal surgery
* Has hemochromatosis, cancer, liver disease, kidney disease, cardiovascular disease, or other coexisting malignancy
* Hemoglobin < 12.5 g/dl (male) or < 11 g/dl (female)
* Severe hypertension (blood pressure > 160/95 mm Hg)
* Has a creatinine greater than 2.0 mg/dl, aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 2 times the upper limit of normal, hematocrit (Hct) less than 32%, or thyroid-stimulating hormone (TSH) less than 0.4 or greater than 5.5 milli-international units (mIU) per liter.
* At the discretion of the study physician or PI, taking medications that affect the outcomes of the study including, but not limited to, corticosteroids, anti-psychotic agents, protease inhibitors, oral contraceptives, estrogens, niacin, and some classes of antidepressants, statins, and antihypertensive medications
* Zinc hypersensitivity
* Use of denture adhesive containing zinc
* Taking other medications or zinc-containing supplements and is unwilling or cannot safely, in the opinion of the study physician, discontinue their use at least 2 weeks prior to protocol initiation
* Any other condition that would, in the opinion of the investigator, place them at an unacceptable risk or render them unable to meet the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Zinc-dependent effect on fasting glucose levels at 1 year | 1 year
  One of the investigator's primary endpoints will be to determine the difference in fasting glucose levels between zinc-treated and placebo-treated individuals after 1 year of receiving study drug
Zinc-dependent effect on HbA1c at 1 year | 1 year
  One of the investigator's primary endpoints will be to determine the difference in HbA1c levels between zinc-treated and placebo-treated individuals after 1 year of receiving study drug

SECONDARY OUTCOMES:
Zinc-dependent effect on fasting glucose levels at 6 months | 6 months
  One of the investigator's secondary endpoints will be to determine the difference in fasting glucose levels between zinc-treated and placebo-treated individuals after 6 months of receiving study drug
Zinc-dependent effect on HbA1c at 6 months | 6 months
  One of the investigator's secondary endpoints will be to determine the difference Hba1c between zinc-treated and placebo-treated individuals after 6 months of receiving study drug

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Lewis, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is possible that deidentified data will be deposited into large public databases as per NIH data sharing policies (e.g. database of Genotypes and Phenotype [dbGAP], Pharmacogenomics Knowledgebase [PharmGKB], etc.). Data to be shared would include, but not limited to, anthropometric data, study outcome data, and relevant covariate data used in statistical models. It is anticipated that data would be available after the completion of the trial. The data will be obtained from the participants and the study-related research procedures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In is anticipated that data would become available following the completion of the study and within 6 months of the publication of the primary analyses.